CLINICAL TRIAL: NCT03273556
Title: Evaluation of the Filler Performance on the Nasolabial Folds of Aliaxin® EV With and Without Lidocaine 0.3%: Comparison Within Subjects (Half Face Method)
Brief Title: Evaluation of the Filler Performance on the Nasolabial Folds of Aliaxin® EV With and Without Lidocaine 0.3%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0817
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Nasolabial Folds Correction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aliaxin® EV Essential Volume (Experimental): Comparison within subjects of Aliaxin® EV Essential Volume with and without Lidocaine 0.3%
  Interventions: Device: Aliaxin® EV Essential Volume (IBSA Farmaceutici Italia S.r.l.) with Lidocaine 0.3%; Device: Aliaxin® EV Essential Volume (IBSA Farmaceutici Italia S.r.l.)

INTERVENTIONS:
Device: Aliaxin® EV Essential Volume (IBSA Farmaceutici Italia S.r.l.) with Lidocaine 0.3% — The injective treatment was performed, during T0 visit after the basal evaluations, mono-laterally on nasolabial fold,(right or left face side in according to a previously defined randomisation list).
  A quantity of Aliaxin® Ev (up to a maximum of 0.5 ml) with Lidocaine 0.3% was injected on the nasolabial fold to achieve the aesthetic correction of the skin defect.
Device: Aliaxin® EV Essential Volume (IBSA Farmaceutici Italia S.r.l.) — The injective treatment was performed on the contralateral nasolabial fold during T0 visit, after the basal evaluations .
  A quantity of Aliaxin® Ev up to a maximum of 0.5 ml was injected on the nasolabial fold to achieve the aesthetic correction of the skin defect.

SUMMARY:
Evaluation of the filler performance on the nasolabial folds of Aliaxin® EV with and without lidocaine 0.3%: comparison within subjects (half face method)

DETAILED DESCRIPTION:
Comparative, randomized, mono-centre spontaneous trial, under dermatological control, that foresaw the comparison within subjects of the investigational product versus investigational product with Lidocaine 0.3% (half face method); assignation of right or left face side to the two injective treatments was choose by the Investigator according to a previously defined randomisation list.

Primary end point of the study was to evaluate the filling and bio-revitalizing activity on nasolabial folds of the product Aliaxin® EV Essential Volume, in women aged 40-65 years.

It was also aim of this study to show if the addition of Lidocaine 0.3% to the investigational product (extemporaneous mixture) could have reduced the discomfort/pain sensation perceived by the subject during the injection procedure, without altering the aesthetic performance.

ELIGIBILITY:
Inclusion Criteria:

* female sex;
* age 40-65 years;
* WSRS 2-4
* asking for nasolabial folds correction;
* execution of any medical/aesthetic procedure, including dental surgery, in the past that foresaw the use of lidocaine as local anesthetic
* available and able to return to the study site for the post-procedural follow-up examinations;
* agreeing to present at each study visit without make-up;
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol or drug abusers;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 (before the aesthetic procedure);
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing skin treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 6 months prior to the study start;
* performing permanent filler in the past;
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 3 months.
* dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne).
* diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy,
* anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago),
* using of drugs able to influence the test results in the investigator opinion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) grade variation from baseline | Baseline visit (T0), Week 4 (T4)
  Reduction of wrinkles severity corresponding to a decrease from the baseline of the Wrinkle Severity Rating Scale (WSRS) clinical score where:
  Grade 1 (absent): no visible nasolabial fold; continuous skin line. Grade 2 (mild): shallow but visible nasolabial fold with a slight indentation; minor facial feature.
  Grade 3 (moderate): moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched.
  Grade 4 (severe): very long and deep nasolabial folds; prominent facial feature; <2mm visible fold when stretched.
  Grade 5 (very severe): extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched.

SECONDARY OUTCOMES:
The Global Aesthetic Improvement Scale (GAIS) grade variation from baseline | Baseline visit (T0), Week 4 (T4)
  Aesthetic improvement in the subjects' midface from their pretreatment state according to a five point scale:
  1. Very much improved: Optimal cosmetic result for the implant in this patient.
  2. Much improved: Marked improvement in appearance from initial condition, but not completely optimal for this patient. A touch up will slightly improve the result.
  3. Improved: Obvious improvement in appearance from the initial condition, but a touch-up or re-treatment is indicated.
  4. No change: The appearance is essentially the same as the original condition.
  5. Worse:The appearance in worst than the original condition.
Self grading | Immediately after the injection procedure (T0A), 2 hours after the injection procedure (T2h)
  Immediately and 2 hours after the aesthetic procedure, each volunteers scored its own sensations thanks to a visual analogic scale (VAS 10 units length) as follow:
  1. Stinging (0= no stinging to 10= strong stinging)
  2. Itching (0= no itching to 10= strong itching)
  3. Tightening (0= no tightening to 10= strong tightening)
  4. Burning (0= no burning to 10= strong burning)
  5. Pain (0= no pain to 10= strong pain)
  6. Discomfort (0= no discomfort to 10= strong discomfort) In order to highlight any differences between the side treated with the investigational product and the one treated with the study product + lidocaine 0.3%, the VAS score will be expressed separately for each of the two treated sides.
Determination of profilometric parameters | Baseline visit (T0), Week 4 (T4)
  Variation from baseline of the nasolabial fold profilometric parameters versus baseline. Profilometric parameters are expressed in in micron.
  A picture of nasolabial fold area is taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to measure skin principal profilometric parameters:Ra (average roughness) Rt (wrinkles total high), Rv (wrinkles maximum depth)

CONTACTS AND LOCATIONS:
Locations (1):
- DermIng S.r.l. Single Member Company, Monza, MB, Italy